CLINICAL TRIAL: NCT02980445
Title: Time Outdoors as an Intervention for Myopia in Children--School-based Randomized Controlled Study
Brief Title: Time Outdoors as an Intervention for Myopia in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEH-M001
Record Dates: First submitted 2016-11-21; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Myopia
Keywords: Myopia; Outdoor time; Children; Intervention; Prevention
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention)
- Outdoor Activity 1 (Experimental): 40min outdoor time in total.
  Interventions: Behavioral: Outdoor activity 1
- Outdoor Activity 2 (Experimental): 80min outdoor time in total
  Interventions: Behavioral: Outdoor activity 2

INTERVENTIONS:
Behavioral: Outdoor activity 1 — 40-minute outdoor activity
  Arms: Outdoor Activity 1
Behavioral: Outdoor activity 2 — Dose 1 plus an additional 40-minute outdoor activities during recesses
  Arms: Outdoor Activity 2

SUMMARY:
The purpose of this study is to determine whether improved outdoor time has an effect on the onset and progression of myopia in children.

DETAILED DESCRIPTION:
1. To evaluate the effect of increased time outdoors on the incidence of myopia in non-myopic children;
2. To evaluate the effect of increased time outdoors on the progression of myopia in myopic children;
3. To explore if there is dose-response effect of time outdoors on the incidence and progression of myopia.

ELIGIBILITY:
Inclusion Criteria:

1. at baseline be enrolled in grade 1 and 2 of primary schools;
2. have a parent or guardian who is able to read and comprehend Mandarin and give informed consent as demonstrated by signing a record of informed consent;
3. Children verbally consent when registration for examination

Exclusion Criteria:

1. Any systemic or ocular pathology that may affect the refractive error status of the eye;
2. Strabismus and amblyopia;
3. Intellectual disability;
4. Using any anti-myopia treatments (orthokeratology, atropine, accommodation function training, acupuncture, auricular point sticking, progressive addition spectacle lenses or other anti-myopia contact lenses).
5. Not suitable for inclusion in the study as deemed by the investigator.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7200 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refractive power（auto-refractor instrument） | 1 year
  The Cycloplegic refraction of all children are measured by auto-refractor(KR-8900, Topcon)

SECONDARY OUTCOMES:
Axial length(IOL Master instrument) | 6 months
  The axial length of the eyeball are measured by IOL Master(version 5.02, Carl Zeiss).

CONTACTS AND LOCATIONS:
Overall Officials: Xun Xu, MD, Principal Investigator — Shanghai Eye Disease Prevention and Treatment Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Sankaridurg P, Naduvilath T, Li W, Morgan IG, Rose KA, Weng R, Xu X, He X. Time outdoors positively associates with academic performance: a school-based study with objective monitoring of outdoor time. BMC Public Health. 2023 Apr 4;23(1):645. doi: 10.1186/s12889-023-15532-y. PMID 37016357
- [Derived] Gong W, Cheng T, Wang J, Zhang B, Chen J, Zhu J, Zou H, Liu K, He X, Xu X. Role of corneal radius of curvature in early identification of fundus tessellation in children with low myopia. Br J Ophthalmol. 2023 Oct;107(10):1532-1537. doi: 10.1136/bjo-2022-321295. Epub 2022 Jul 26. PMID 35882514
- [Derived] He X, Sankaridurg P, Wang J, Chen J, Naduvilath T, He M, Zhu Z, Li W, Morgan IG, Xiong S, Zhu J, Zou H, Rose KA, Zhang B, Weng R, Resnikoff S, Xu X. Time Outdoors in Reducing Myopia: A School-Based Cluster Randomized Trial with Objective Monitoring of Outdoor Time and Light Intensity. Ophthalmology. 2022 Nov;129(11):1245-1254. doi: 10.1016/j.ophtha.2022.06.024. Epub 2022 Jun 30. PMID 35779695